CLINICAL TRIAL: NCT03350893
Title: Efficacy Evaluation of the Probiotics Containing Skincare Products on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Chia Nan University of Pharmacy and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-047-A2
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Skin Problems
MeSH Terms: interventions — Probiotics; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel, Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Emulsion base without probiotics
  Interventions: Other: Emulsion base
- Active Group (Experimental): Emulsion base with probiotics
  Interventions: Combination Product: Emulsion base with probiotics

INTERVENTIONS:
Combination Product: Emulsion base with probiotics — Water、Polyglyceryl-3/ Methylglucose Distearate、Triethyl Hexanoin、Macadamia Ternifolia Seed Oil、Propanediol、PEG/PPG/Polybutylene Glycol-8/5/3 Glycerin、Cetyl Alcohol、Myristyl Myristate、Glycerin、Glycosyl Trehalose/Hydrogenated Starch Hydrolysate、Rice Ferment Filtrate(Sake)、Saccharomyces/Daylily Flower Ferment Filtrate、Bis-PEG/PPG-20/5 PEG/PPG-20/5Dimethicone、Methoxy PEG/PPG-25/4 Dimethicone、Caprylic/Capric Triglyceride、Sodium Polyacrylate、Phenoxyethanol、o-Cymen-5-ol、Xanthan Gum、Potassium Hydroxide, Heat-killed L. plantarum powders (1x10^9 cells/ g-cream)
  Other Names: Active Group
  Arms: Active Group
Other: Emulsion base — Water、Polyglyceryl-3/ Methylglucose Distearate、Triethyl Hexanoin、Macadamia Ternifolia Seed Oil、Propanediol、PEG/PPG/Polybutylene Glycol-8/5/3 Glycerin、Cetyl Alcohol、Myristyl Myristate、Glycerin、Glycosyl Trehalose/Hydrogenated Starch Hydrolysate、Rice Ferment Filtrate(Sake)、Saccharomyces/Daylily Flower Ferment Filtrate、Bis-PEG/PPG-20/5 PEG/PPG-20/5Dimethicone、Methoxy PEG/PPG-25/4 Dimethicone、Caprylic/Capric Triglyceride、Sodium Polyacrylate、Phenoxyethanol、o-Cymen-5-ol、Xanthan Gum、Potassium Hydroxide
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
Previous studies on skin health with Lactic acid bacteria (LAB) have been published for many years, including prevention of skin diseases and improvement of skin conditions. In this clinical study, the investigators researched the benefit effects of heat-killed Lactobacillus plantarum cream on skin health.

DETAILED DESCRIPTION:
To evaluate the efficacy of applying probiotic cream in the ameliorationof the whole face skin conditions such as moisturizing, whitening, anti-wrinkle and so on.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 20-60.

Exclusion Criteria:

* Subjects with photosensitivity (Sun allergy).
* Subjects are undergoing medical therapy for skin diseases.
* Subjects with severe hyperpigmentation.
* Subjects with diabetes.
* Subjects with cosmetics allergy.
* Subjects who have recently participated laser therapies or other treatments are not suitable for sun.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Skin Diagnosis | Baseline, 4 weeks and 8 weeks
  The changes of skin condition by VISIA Complexion Analysis System

SECONDARY OUTCOMES:
Skin Moisture | Baseline, 4 weeks and 8 weeks
  The changes of skin moisture by Skicon-200EX and Corneometer CM 825
Skin Color | Baseline, 4 weeks and 8 weeks
  The changes of skin color by DermaSpectrometer

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Gong Lin, PhD, Study Chair — Chia Nan University of Pharmacy and Science, Taiwan, R.O.C.
Locations (1):
- Chia Nan University of Pharmacy and Science, Tainan, Taiwan